CLINICAL TRIAL: NCT05760508
Title: Novel Markers of Disease Progression in Interstitial Lung Disease
Acronym: NOMAD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, RICHELDI LUCA, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 2104
Record Dates: First submitted 2023-02-10; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study design: A prospective cohort study with a longitudinal design, with several parameters measured serially at baseline and at pre-specified time points during three to five years of clinical observation.

Primary objective: To validate quantitative analysis of lung sounds as a marker of disease progression in a cohort of patients with Interstitial Lung Disease (ILD) via correlation with the extent of fibrosis on HRCT, measured both via visual scoring and quantitative CT assessment, and other validated parameters of disease progression such as FVC, tolerance to exercise and patient-related outcomes (symptoms and quality of life).

Secondary objectives: To determine the prognostic value of quantitative analysis of lung sounds and a series of novel putative biological markers, obtained from peripheral blood and bronchoalveolar lavage, toward poor outcomes (death, categorical decline of % predicted FVC >10%, acute exacerbation or respiratory-related hospitalisations) as compared to more conventional clinical, physiology and radiologic measurements.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of ILD, made according to international guidelines where available
* age between 40 and 90 years

Exclusion Criteria:

* significant comorbidities or physical impairment that could affect participation

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with a diagnosis of ILD
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Disease progression | 3 years
  Validate quantitative analysis of lung sounds as a marker of disease progression via correlation with the extent of fibrosis on HRCT, measured both via visual scoring and quantitative CT assessment, and other validated parameters of disease progression such as FVC, tolerance to exercise and patient-related outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Agostino Gemelli IRCCS, Rome, Roma, Italy